CLINICAL TRIAL: NCT01164709
Title: Phase I Trial of Nelfinavir and Bortezomib in Advanced Hematologic Malignancies
Brief Title: Nelfinavir Mesylate and Bortezomib in Treating Patients With Relapsed or Progressive Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 65/08; SWS-SAKK-65/08; EU-21051; SWS-SAKK-JC26866138LYM1005; CDR0000681442 (Registry Identifier: CDR0000681442)
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Leukemia; Lymphoma; Mature T-cell and Nk-cell Neoplasms; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent mantle cell lymphoma; recurrent adult T-cell leukemia/lymphoma; adult nasal type extranodal NK/T-cell lymphoma; angioimmunoblastic T-cell lymphoma; peripheral T-cell lymphoma; T-cell large granular lymphocyte leukemia; anaplastic large cell lymphoma; recurrent grade 3 follicular lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; aggressive NK-cell leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma, Mantle-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Leukemia, Large Granular Lymphocytic; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Follicular; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Congenital Abnormalities; Leukemia, Prolymphocytic | interventions — Bortezomib; Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bortezomib + nelfinavir (Experimental): escalation 3 by 3 cohorts
  Interventions: Drug: bortezomib; Drug: nelfinavir mesylate

INTERVENTIONS:
Drug: bortezomib — Bortezomib i.v., day 8, 11, 15, 18; 1.3 mg/m2
  Other Names: Velcade
Drug: nelfinavir mesylate — p.o., days 1 to 21; dose level: (625), 1250, 1875, or 2500 mg, 2x/d
  Other Names: Viracept

SUMMARY:
RATIONALE: Nelfinavir mesylate and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bortezomib may also stop the growth of hematologic cancer by blocking blood flow to the cancer. Giving nelfinavir mesylate together with bortezomib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of nelfinavir mesylate when given together with bortezomib in treating patients with relapsed or progressive advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the safety of nelfinavir mesylate in combination with bortezomib in patients with relapsed or progressive, advanced hematologic malignancies.
* To establish the phase II recommended dose of nelfinavir mesylate in these patients.

OUTLINE: This is a multicenter, dose-escalation study of nelfinavir mesylate.

Patients receive oral nelfinavir mesylate twice daily on days 1-21 and bortezomib IV on days 8, 11, 15, and 18 in course 1. Course 1 has a duration of 28 days. Beginning in course 2, patients receive oral nelfinavir mesylate twice daily on days 1-14 and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for 2 courses. Patients with responding disease may continue to receive nelfinavir mesylate and bortezomib for up to 4 additional courses.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with advanced hematologic malignancies meeting the following criteria:

  * Multiple myeloma

    * Received ≥ 2 lines of prior chemotherapy (induction chemotherapy followed by high-dose chemotherapy and autologous stem cell transplant with or without maintenance therapy is considered one line of therapy)
  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Diffuse large B-cell lymphoma
  * Hodgkin lymphoma
  * Mantle cell lymphoma
  * Mature T- and NK-cell neoplasms restricted to the following WHO-defined entities:

    * T-cell prolymphocytic leukemia
    * T-cell large granular lymphocytic leukemia
    * Aggressive NK-cell leukemia
    * Adult T-cell leukemia/lymphoma
    * Extranodal NK/T-cell lymphoma (nasal type)
    * Mycosis fungoides
    * Sézary syndrome
    * Primary CD30-positive T-cell lymphoproliferative disorders
    * Primary cutaneous anaplastic large cell lymphoma
    * Primary cutaneous gamma-delta T-cell lymphoma
    * Peripheral T-cell lymphoma (not otherwise specified)
    * Angioimmunoblastic T-cell lymphoma
    * Anaplastic large cell lymphoma (ALK-positive/ALK-negative)
  * Grade 3B follicular lymphoma
* Relapsed following or progressed during standard therapy
* Meeting the following criteria:

  * Standard intensive therapy is not feasible
  * Current disease state for which there is no standard effective therapy
  * Refused standard therapy where no curative option exists
* Measurable disease, defined as the following:

  * Myeloma: measurable serum monoclonal protein > 1 g/dL for IgG, or > 0.5 g/dL for IgA, IgM or IgD, or difference between involved and uninvolved free light chain levels in serum > 100 mg/L
  * Lymphoma: must have ≥ 1 lesion measurable by CT (longest diameter ≥ 15 mm)
  * Acute leukemia: ≥ 20% blasts in bone marrow or in peripheral blood (≥ 200/mL blasts in peripheral blood)
* No HIV-associated lymphoma

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³ (if bone marrow impairment, ≥ 20,000/mm^3)
* Hemoglobin > 80 g/L (if considered to be caused by the underlying hematologic malignancy or bone marrow impairment, > 80 g/L after transfusion)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (if suspected hemolysis, direct bilirubin ≤ 1.5 times ULN)
* ALT ≤ 2.5 times ULN
* Calculated creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Willing and capable to comply with an oral regimen
* Capable of understanding information given by the investigator on the trial
* Able to adhere and remain in geographic proximity to allow proper staging, treatment, and followup
* No other non-hematologic malignancy within the past 5 years, except adequately treated cervical carcinoma in situ or localized nonmelanoma skin cancer
* No known chronic hepatitis B or C infection or known HIV infection
* No serious underlying medical condition (at the judgment of the investigator) which would impair the ability of the patient to participate in the trial, including any of the following:

  * Active autoimmune disease
  * Uncontrolled diabetes
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric disorder
* No myocardial infarction within the past 6 months
* No polyneuropathy > grade 1 significantly interfering with activities of daily living or painful polyneuropathy
* No known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 4 prior lines of chemotherapeutic regimens (induction chemotherapy followed by high-dose chemotherapy and autologous stem cell transplant with or without maintenance therapy is considered one line of therapy)
* More than 30 days since prior treatment in a clinical trial
* More than 30 days since prior and no concurrent chemotherapy or biologic agents

  * For patients with acute leukemia, hydroxyurea may be given up to 48 hours before first administration of the trial treatment, and low dose cytarabine (up to 20 mg/m^2) and mitoxantrone up to 20 mg up to 14 days before first dosing
* At least 1 week since prior and no concurrent CYP3A4 modulators
* No concurrent other experimental drugs
* No concurrent radiotherapy
* No concurrent antineoplastic therapy with chemotherapeutic or biologic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | during first cycle

SECONDARY OUTCOMES:
Objective response | during treatment
Adverse events according to NCI CTCAE v.4.0 | during treatment + 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Driessen, MD, Study Chair — Cantonal Hospital of St. Gallen; Dagmar Hess, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Roger von Moos, MD, Principal Investigator — Kantonsspital Graubuenden; Thomas Pabst, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (4):
- Switzerland (4):
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Result] Driessen C, Kraus M, Joerger M, Rosing H, Bader J, Hitz F, Berset C, Xyrafas A, Hawle H, Berthod G, Overkleeft HS, Sessa C, Huitema A, Pabst T, von Moos R, Hess D, Mey UJ. Treatment with the HIV protease inhibitor nelfinavir triggers the unfolded protein response and may overcome proteasome inhibitor resistance of multiple myeloma in combination with bortezomib: a phase I trial (SAKK 65/08). Haematologica. 2016 Mar;101(3):346-55. doi: 10.3324/haematol.2015.135780. Epub 2015 Dec 11. PMID 26659919